CLINICAL TRIAL: NCT03136588
Title: The Efficacy and Stability of Information and Communication Technology Based Centralized Clinical Trial Monitoring System of Adherence to Immunosuppressive Medication in Kidney Transplant Recipients
Brief Title: Information and Communication Technology (ICT) Based Centralized Clinical Trial Monitoring System for Drug Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy, Republic of Korea (Other Government); Korea Evaluation Institute of Industrial Technology (Other); Daegu Metropolitan City, Korea (Other Government); ICT Clinical Trial Coordination Center (Other)
Responsible Party: Principal Investigator, Yong-Lim Kim, Principal Investigator, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICT_COM_P01_KT-ver2.4
Record Dates: First submitted 2017-04-20; First posted 2017-05-02 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Kidney Transplantation
Keywords: Information and Communication Technology; Adherence; Kidney transplantation

STUDY DESIGN:
Intervention Model Description: randomized in a 1:1 ratio to either Information and Communication Technology (ICT) based centralized clinical trial monitoring system or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICT based monitoring group (Experimental): Intervention: In the ICT-based centralized monitoring group, both subjects and medical staff receive feedbacks regarding a missed dose, misuse, and overuse of the medication in the form of text messages and pill box alarms.
  Interventions: Device: Feedback using ICT based monitoring system
- Control group (No Intervention): Use standard questionnaire to gather information for drug adherence

INTERVENTIONS:
Device: Feedback using ICT based monitoring system — In case of a missed immunosuppressant dose, the first violation does not generate a feedback while the second one does within one hour at the break of the ±3 hour range from the fixed dosing time. Up to two additional alarms/texts are sent at an interval of 30 minutes if the dose is still not taken after the feedback. For any discrepancy between the dosage taken and the dosage prescribed, a feedback is sent within 1 hour from the moment of recognition. Again, the first violation goes without response, while any violation after that generates feedbacks. Similarly, if a dose is taken outside of the allowed ±3 hour dosing time range, a feedback is sent within 1 hour of recognition, starting with the second violation.
  Arms: ICT based monitoring group

SUMMARY:
Immunosuppression non-adherence in kidney transplant recipients (KTRs) not only increases the risk of medical intervention due to acute rejection and graft loss but burdens the socioeconomic system in the form of increased healthcare cost. Aggressive preemptive effort by healthcare professionals geared to ensure adherence to immunosuppressants in KTRs is significant and imperative.

This study was designed as a prospective, randomized, controlled, and multicenter study aimed at evaluating efficacy and stability of the information and communication technology (ICT)-based centralized monitoring system in boosting medication adherence in KTRs.

This study is based upon work supported by the Ministry of Trade, Industry & Energy (MOTIE, Korea) under Industrial Technology Innovation Program ( No. 10059066, 'Establishment of ICT Clinical Trial System and Foundation for Industrialization').

DETAILED DESCRIPTION:
This study has a multi-center, open-label, prospective, and randomized clinical trial design. One hundred KTRs who fill out the informed consent form are registered and randomized 1:1 into the ICT-based centralized clinical trial monitoring group (n=50) or the ambulatory follow-up group (n=50). The planned follow-up duration is 6 months. The ICT-based centralized clinical trial monitoring group is given a smart pill box equipped with personal identification system. Fingerprint registration is required in advance, so that it would be used for authentication before each use of the smart pill box later. The adherence-related information obtained from the pill box is saved, monitored, and sent out via a home-monitoring system. In the ICT-based centralized clinical trial monitoring group, feedback is sent to both patients and medical staff in the form of texts and pill box alarms if there is a dosage/dosing time error or a missed dose.

Both groups are to make 6 office visits after randomization at 4, 8, 12, 16, 20, and 24 weeks. Each visit requires measurement of blood drug level, creatinine level, and estimated glomerular filtration rate. Serum BK virus is assessed at 12 weeks, and panel reactive antibody at 24 weeks. Both groups keep a drug administration diary that specifies date, a dose taken or not, dosing time, and dosage. At each visit, subjects go over the diary with investigators and fill out a questionnaire using the Modified Morisky Scale. The ICT-based centralized clinical trial monitoring group completes a patient satisfaction questionnaire developed by the ICT clinical trial support center at 4 and 12 weeks.

The objective of this study is

1. to evaluate the effectiveness of ICT based centralized clinical trial monitoring system on adherence of immunosuppressive agents
2. to study the influence of ICT based centralized monitoring on immunosuppressive and clinical outcomes including therapeutic trough level
3. to evaluate patient's satisfaction about ICT based clinical trial monitoring system

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 19 and over
2. At least 1 month lapsing from kidney transplantation
3. Stable renal function maintained after kidney transplantation(eGFR ≥ 30 mL/min/1.73m2)
4. History of kidney transplantation only and no other organs
5. Use of tacrolimus, mycophenolic acid, and steroids for post-transplant immunosuppression
6. Patients, with capability and willingness to give consent to trial participation, who have signed the informed consent form in compliance with due process and are capable of making office visits and taking part in the trial as required by the protocol.

Exclusion Criteria:

1. Patients' refusal of the ICT-based centralized home monitoring
2. History of treatment for acute rejection within the past 3 months
3. Active infectious disease
4. Uncorrected ischemic heart disease
5. Visual or auditory defects that could affect use of the smart pill box
6. Fingerprint authentication of personal identity deemed impossible (ex: adermatoglyphia)
7. Other reasons determined by investigators that make participation in the clinical trial inappropriate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Drug adherence | at 6 months after enrollment
  To evaluate the effectiveness of ICT based clinical trial monitoring system on the compliance of immunosuppressive medications.

SECONDARY OUTCOMES:
Immunosuppressive drug levels | At every 4 weeks up to 24 weeks after enrollment
  Tacrolimus, Mycophenolic acid trough level
Incidence of biopsy-proven acute rejection | Up to 24 weeks after enrollment
  Biopsy-proven acute rejection
Development of de novo panel reactive antibody | Up to 24 weeks after enrollment
  De novo panel reactive antibody
Development of polyomavirus (BK virus) infection | Up to 24 weeks after enrollment
  Polymerase chain reaction (PCR) of blood BK virus
Changes in renal allograft function | From baseline to 24 weeks after enrollment
  Serum creatinine, estimated glomerular filtration rate
Changes in ICT-based centralized monitoring system satisfaction scores of patients assessed by system satisfaction questionnaire | From 4 weeks to 24 weeks after enrollment
  System satisfaction questionnaire score
Malfunction rate of ICT-based centralized monitoring system | Up to 24 weeks after enrollment
  Malfunction rate

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Lim KIM, MD, PhD, Principal Investigator — Kyungpook National University Hospital
Locations (2):
- South Korea (2):
  - Konyang University Hospital, Daejeon
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sellares J, de Freitas DG, Mengel M, Reeve J, Einecke G, Sis B, Hidalgo LG, Famulski K, Matas A, Halloran PF. Understanding the causes of kidney transplant failure: the dominant role of antibody-mediated rejection and nonadherence. Am J Transplant. 2012 Feb;12(2):388-99. doi: 10.1111/j.1600-6143.2011.03840.x. Epub 2011 Nov 14. PMID 22081892
- [Background] Pinsky BW, Takemoto SK, Lentine KL, Burroughs TE, Schnitzler MA, Salvalaggio PR. Transplant outcomes and economic costs associated with patient noncompliance to immunosuppression. Am J Transplant. 2009 Nov;9(11):2597-606. doi: 10.1111/j.1600-6143.2009.02798.x. PMID 19843035
- [Background] Schafer-Keller P, Steiger J, Bock A, Denhaerynck K, De Geest S. Diagnostic accuracy of measurement methods to assess non-adherence to immunosuppressive drugs in kidney transplant recipients. Am J Transplant. 2008 Mar;8(3):616-26. doi: 10.1111/j.1600-6143.2007.02127.x. PMID 18294158
- [Background] Claxton AJ, Cramer J, Pierce C. A systematic review of the associations between dose regimens and medication compliance. Clin Ther. 2001 Aug;23(8):1296-310. doi: 10.1016/s0149-2918(01)80109-0. PMID 11558866
- [Background] Henriksson J, Tyden G, Hoijer J, Wadstrom J. A Prospective Randomized Trial on the Effect of Using an Electronic Monitoring Drug Dispensing Device to Improve Adherence and Compliance. Transplantation. 2016 Jan;100(1):203-9. doi: 10.1097/TP.0000000000000971. PMID 26588006
- [Background] Christensen A, Christrup LL, Fabricius PE, Chrostowska M, Wronka M, Narkiewicz K, Hansen EH. The impact of an electronic monitoring and reminder device on patient compliance with antihypertensive therapy: a randomized controlled trial. J Hypertens. 2010 Jan;28(1):194-200. doi: 10.1097/HJH.0b013e328331b718. PMID 19770778
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Jung HY, Jeon Y, Seong SJ, Seo JJ, Choi JY, Cho JH, Park SH, Kim CD, Yoon YR, Yoon SH, Lee JS, Kim YL. ICT-based adherence monitoring in kidney transplant recipients: a randomized controlled trial. BMC Med Inform Decis Mak. 2020 Jun 10;20(1):105. doi: 10.1186/s12911-020-01146-6. PMID 32522263
- [Derived] Jung HY, Seong SJ, Choi JY, Cho JH, Park SH, Kim CD, Yoon YR, Kim HK, Huh S, Yoon SH, Lee JS, Kim YL. The efficacy and stability of an information and communication technology-based centralized monitoring system of adherence to immunosuppressive medication in kidney transplant recipients: study protocol for a randomized controlled trial. Trials. 2017 Oct 16;18(1):480. doi: 10.1186/s13063-017-2221-z. PMID 29037222